CLINICAL TRIAL: NCT01354522
Title: A Randomized, Phase III Study Comparing TAC (Docetaxel, Doxorubicin, Cyclophosphamide) With TCX ( Docetaxel, Cyclophosphamide, Capecitabine) as Adjuvant Treatment for High-risk Her2-Negative Breast Cancer
Brief Title: TAC Versus TCX as Adjuvant Treatment for High-risk Her2-Negative Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-Breast-TCX
Record Dates: First submitted 2011-05-09; First posted 2011-05-17 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2014-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Doxorubicin; Cyclophosphamide; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | US Export: No

ARMS (2):
- TAC (Active Comparator): docetaxel 75 mg/m², iv, day 1 doxorubicin 50 mg/m² or epirubicin 75mg/m², iv, day 1 Cyclophosphamide 500 mg/m², iv, day 1 every 3 weeks for 6 cycles
  Interventions: Drug: Docetaxel, Doxorubicin, Cyclophosphamide
- TCX (Experimental): docetaxel 75 mg/m², iv, day 1 Cyclophosphamide 500 mg/m², iv, day 1 capecitabine 950 mg/m2, twice a day, via oral intake, day 1 to day 14 every 3 weeks for 6 cycles
  Interventions: Drug: Docetaxel, Cyclophosphamide, Capecitabine

INTERVENTIONS:
Drug: Docetaxel, Doxorubicin, Cyclophosphamide — docetaxel 75 mg/m², iv, day 1 doxorubicin 50 mg/m² or epirubicin 75mg/m², iv, day 1 Cyclophosphamide 500 mg/m², iv, day 1 every 3 weeks for 6 cycles
  Arms: TAC
Drug: Docetaxel, Cyclophosphamide, Capecitabine — docetaxel 75 mg/m², iv, day 1 Cyclophosphamide 500 mg/m², iv, day 1 capecitabine 950 mg/m2, twice a day, via oral intake, day 1 to day 14 every 3 weeks for 6 cycles
  Arms: TCX

SUMMARY:
Some sub-analysis has shown anthracycline-based regimens are not effective in Her-2 negative breast cancer, while capecitabine is more effective in this group of patients.

This is a prospective, randomised phase III trial, to compare the efficacy and safety profiles of two types of adjuvant chemotherapy regimens for HER2 negative, node positive or node-negative high-risk breast cancer patients.

Control Arm: This includes 6 cycles of TAC 75/50/500 mg/m2 day 1 every 3 weeks. Experimental Arm: This includes 6 cycles of TC 75/500 mg/m2, day 1 every 3 weeks, concurrently with capecitabine 950 mg/m2, twice a day, via oral intake, for 14 days, and then a one-week rest period.

Women with hormone receptor positive tumours must receive 5 years endocrine after the end of chemotherapy.

Patients may receive radiotherapy when clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Histological diagnosis of operable invasive adenocarcinoma of the breast (T1-T3). Tumours must be HER2 negative. Time window between surgery and study randomization must be less than 60 days.
* Surgery must consist of mastectomy or conservative surgery with axillary lymph node dissection. Margins free of disease and ductal carcinomas in situ (DCIS) are required. Lobular carcinoma is not considered a positive margin.
* Positive axillary lymph nodes defined as at least 1 out of 10 nodes with presence of disease. If sentinel node technique is used, sentinel node can be the only node affected.
* Node-negative high-risk breast cancer was defined as tumors with a size ≥ 2 cm, fulfilling at least one of the following criteria: histological grade 3, estrogen receptor (ER)-negative and progesterone receptor (PR)-negative, or a Ki67 proliferation index ≥ 14%.
* Status of hormone receptors in primary tumour. Results must be available before the end of adjuvant chemotherapy.
* Patients must not present evidence of metastatic disease. Status of HER2 in primary tumour, known before randomization. Patients with immune histochemistry (IHC) 0 or +1 are eligible. For patients with ICH 2+, fluorescence in situ hybridization (FISH) is mandatory and result must be negative.
* Age >= 18 and <= 70 years old.
* Performance status (Karnofsky index) >= 70.
* Normal electrocardiogram (EKG) in the 12 weeks prior to randomization. If needed, normal cardiac function must be confirmed by left ventricular ejection fraction (LVEF).
* Laboratory results (within 14 days prior to randomization):

  * Hematology: neutrophils >= 1.5 x 10^9/l; platelets >= 100 x 10^9/l; hemoglobin >= 10 mg/dl;
  * Hepatic function: total bilirubin <= 1 upper normal limit (UNL); SGOT and SGPT <= 2.5 UNL; alkaline phosphatase <= 2.5 UNL. If values of SGOT and SGPT > 1.5 UNL are associated to alkaline phosphatase > 2.5 UNL, patient is not eligible;
  * Renal function: creatinine <= 175 mmol/l (2 mg/dl); creatinine clearance >= 60 ml/min;
* Complete stage workup during the 12 weeks prior to randomization (mammograms are allowed within a 20 week window). All patients must have a bilateral mammogram, thorax x-ray, abdominal echography and/or computed tomography (CT)-scan. If bone pain, and/or alkaline phosphatase elevation, a bone scintigraphy is mandatory. This test is recommended for all patients. Other tests: as clinically indicated.
* Patients able to comply with treatment and study follow-up.
* Negative pregnancy test done in the 14 prior days to randomization.

Exclusion Criteria:

* Prior systemic therapy for breast cancer.
* Prior therapy with anthracyclines or taxanes (paclitaxel or docetaxel) for any malignancy.
* Prior radiotherapy for breast cancer.
* Bilateral invasive breast cancer.
* Pregnant or lactating women. Adequate contraceptive methods must be used during chemotherapy and hormone therapy treatments.
* Any T4 or M1 tumour.
* HER2 positive breast cancer (IHC 3+ or positive FISH result).
* Pre-existing grade >= 2 motor or sensorial neurotoxicity (National Cancer Institute Common Toxicity Criteria version 2.0 [NCI CTC v-2.0]).
* Any other serious medical pathology, such as congestive heart failure; unstable angina; history of myocardial infarction during the previous year; uncontrolled HA or high risk arrhythmias.
* History of neurological or psychiatric disorders, which could preclude the patients from free informed consent.
* Active uncontrolled infection.
* Active peptic ulcer; unstable diabetes mellitus.
* Previous or current history of neoplasms different from breast cancer, except for skin carcinoma, cervical in situ carcinoma, or any other tumour curatively treated and without recurrence in the last 10 years; ductal in situ carcinoma in the same breast; lobular in situ carcinoma.
* Chronic treatment with corticosteroids.
* Contraindications for corticosteroid administration.
* Concomitant treatment with raloxifene, tamoxifen or other selective estrogen receptor modulators (SERMs), either for osteoporosis treatment or for prevention. These treatments must stop before randomisation.
* Concomitant treatment with other investigational products; participation in other clinical trials with a non-marketed drug in the 20 previous days before randomization.
* Concomitant treatment with another therapy for cancer.
* Males.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 10 years
  the time from the date of surgery to locoregional or distant recurrence, second primary malignancy or death, whichever occurred first
overall survival | 10 years
  the time from the date of surgery to the date of death from any cause

SECONDARY OUTCOMES:
distant disease-free survival | 10 years
  the time from randomization to distant recurrence of breast cancer
Adverse event rate (CTCAE v. 4.0) | 10 years
disease-specific survival | 10 years
  the time from randomization to deaths caused by breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Sun, Master, Study Chair — PUMCH
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Song Y, Wang Y, Cao X, Xu Y, Zhou Y, Sun Q, Shen S. Adjuvant capecitabine in combination with docetaxel and cyclophosphamide versus anthracycline plus docetaxel and cyclophosphamide regimen in women with high-risk, HER2-negative breast cancer: An open-label, randomized controlled trial. Cancer Commun (Lond). 2025 Sep;45(9):1113-1122. doi: 10.1002/cac2.70041. Epub 2025 Jun 9. PMID 40491042
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241